CLINICAL TRIAL: NCT05495217
Title: A Single-center, Randomized, Controlled Clinical Study for Comparison of the Effects Between Gasless Laparoscopy-assisted and Conventional Laparoscopy-assisted Gastrectomy With D2 Lymphadenectomy for Distal Gastric Cancer
Brief Title: A Clinical Study for Comparison of the Effects Between Gasless Laparoscopy and Conventional Laparoscopy for Distal Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xue Yingwei (Other)
Responsible Party: Sponsor-Investigator, Xue Yingwei, Director, Head of Gastrointestinal surgery, Principal Investigator, Clinical Professor, The Third Affiliated Hospital of Harbin Medical University
Organization: The Third Affiliated Hospital of Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJS2021-13
Record Dates: First submitted 2022-07-23; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Gastrectomy; Laparoscopy
Keywords: Laparoscopy-assisted Gastrectomy; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gasless Laparoscopy-assisted Gastrectomy (Experimental): Patients receive Gasless Laparoscopy-assisted Gastrectomy with D2 Lymphadenectomy for Distal Gastric Cancer.
  Interventions: Device: Gasless Laparoscopy
- Conventional Laparoscopy-assisted Gastrectomy (Other): Patients receive Conventional Laparoscopy-assisted Gastrectomy with D2 Lymphadenectomy for Distal Gastric Cancer.
  Interventions: Device: Conventional Laparoscopy

INTERVENTIONS:
Device: Conventional Laparoscopy — A procedure in which a laparoscope (LAPAROSCOPES) is inserted through a small incision near the navel to examine the abdominal and pelvic organs in the PERITONEAL CAVITY using Induced pneumoperitoneum.
  Other Names: Laparoscopic Surgery
  Arms: Conventional Laparoscopy-assisted Gastrectomy
Device: Gasless Laparoscopy — A procedure in which a laparoscope (LAPAROSCOPES) is inserted through a small incision near the navel to examine the abdominal and pelvic organs in the PERITONEAL CAVITY without Induced pneumoperitoneum.It mechanically elevates the abdominal wall and allows laparoscopic visualization through a single incision, providing diagnostic and therapeutic procedures.
  Other Names: Gasless Laparoscopic Surgery
  Arms: Gasless Laparoscopy-assisted Gastrectomy

SUMMARY:
The aim of this trial is to confirm the non-inferiority of Gasless laparoscopy-assisted distal D2 radical gastrectomy to the conventional laparoscopy-assisted distal D2 radical gastrectomy for the treatment of advanced gastric cancer patients (T2-4a, N0-3, M0).

DETAILED DESCRIPTION:
The primary end point was operative time for Gasless laparoscopy-assisted distal D2 radical gastrectomy and conventional laparoscopy-assisted distal D2 radical gastrectomy. The secondary outcomes of interest were intraoperative vital signs; postoperative pain; and surgeon satisfaction for D2 radical gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <75 years old;
2. The gastric primary lesion is diagnosed as gastric adenocarcinoma by endoscopic biopsy histopathologic techniques (papillary adenocarcinoma [pap], tubular adenocarcinoma [tub], mucinous adenocarcinoma [muc], signet ring cell carcinoma [sig], and poorly differentiated adenocarcinoma [por]);
3. Preoperative clinical staging of T2-4a, N0-3, M0 (see preoperative assessment program; tumor staging is in accordance with AJCC-7th TNM);
4. It is expected that R0 surgical results will be obtained by distal subtotal gastrectomy and D2 lymph node dissection (also applies to multiple primary tumors)
5. Preoperative ECOG status score of 0/1;
6. Preoperative ASA (American society of anesthesiology) class of I -III;
7. Patients signed informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Serious mental illness;
3. History of abdominal surgery (except for laparoscopic cholecystectomy);
4. History of gastric surgery (including ESD/EMR for gastric cancer);
5. Preoperative imaging examination suggests regional integration enlargement of lymph nodes (maximum diameter ≥3 cm)
6. Other malignant disease history within five (5) years;
7. Patients who received or were recommended a new adjuvant therapy;
8. History of unstable angina or myocardial infarction within six (6) months;
9. History of cerebral infarction or cerebral hemorrhage within six (6) months;
10. History of sustained systemic corticosteroid therapy within one (1) month;
11. Patients requiring simultaneous surgical treatment of other diseases;
12. Gastric cancer complications (bleeding, perforation, obstruction) requiring emergency surgery;
13. Pulmonary function test with FEV1 <50% of the expected value.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | During procedure.
  The primary end point was operative time for Gasless Laparoscopy-assisted Gastrectomy with D2 Lymphadenectomy and conventional Laparoscopy-assisted Gastrectomy with D2 Lymphadenectomy.

SECONDARY OUTCOMES:
Blood pressure | Through study completion, an average of 2 year.
  Intraoperative blood pressure
End-tidal carbon dioxide | Through study completion, an average of 2 year.
  Intraoperative end-tidal carbon dioxide
Heart rate | Through study completion, an average of 2 year.
  Intraoperative heart rate
Estimated blood loss | Through study completion, an average of 2 year.
  Intraoperative estimated blood loss
Complications | Through study completion, an average of 2 year.
  Intraoperative complications
Death | Through study completion, an average of 2 year.
  Intraoperative death
Blood transfusion | Through study completion, an average of 2 year.
  Intraoperative and postoperative blood transfusion
Tumor size | Through study completion, an average of 2 year.
  Tumor size

CONTACTS AND LOCATIONS:
Overall Officials: Yingwei Xue, doctor, Study Director — Harbin Medical University
Locations (1):
- Harbin University Cancer Hospital, Harbin, Heilongjiang, China